CLINICAL TRIAL: NCT01416857
Title: ED Disability Diagnostic Tool: a Health Information Technology Feasibility Study
Brief Title: Emergency Department (ED) Disability Diagnostic Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1004006652; 1R01 HS0184120-01A1
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Disability Diagnosis
Keywords: Medicare

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOD (No Intervention): Group evaluated using the currently available ED measure of disability (MOD)
- RDDT (Experimental): Group will be evaluated using ED Rasch Disability Diagnostic Tool (RDDT)
  Interventions: Other: RDDT

INTERVENTIONS:
Other: RDDT
  Arms: RDDT

SUMMARY:
Aim 1: To develop and validate an Emergency Department(ED) Rasch Disability Diagnostic Tool (RDDT).

Hypothesis:

* Rasch modeling will provide an instrument with better measurement properties, including increased reliability and validity compared to currently available ED measure of disability (MOD).

Aim 2: To conduct a randomized controlled trial to evaluate the utility of the ED-RDDT to reduce rehospitalizations in Medicare recipients visiting an urban Emergency Department for non-traumatic illness

Hypotheses:

* Compared to the standard screening tool, the ED RDDT will reduce reutilization of the hospital (ED visits, hospital admissions, or death) within 60 days of discharge.
* The ED RDDT will reduce costs to Medicare, hospitals and patients.

DETAILED DESCRIPTION:
Research Overview - The overarching aim of this study is to improve health outcomes for patients presenting to EDs by modifying and testing a disability diagnostic tool. The investigators expect a more accurate and precise tool will lead to better discharge plans and referrals for ED patients, reduce morbidity and mortality, and reduce unnecessary hospital visits and costs. The investigators will develop the core set of indicators with face (logical) validity from our research team of disability, emergency medicine, and geriatric medicine experts and practitioners. These experts will choose which pieces of information need to be included and group the selected pieces of information into content areas. Each content area will contain pieces of information that measure the same unidimensional concept. The investigators go through a series of Rasch analyses to establish which sets of information are in fact unidimensional and form usable scales. The investigators will test the validity of this preliminary version of the RDDT on existing hospital data by using it to predict health outcomes. Finally the investigators will consult the panel of experts to determine which information items, if any, are essential and missing from each content area. If there are such items they will be added to the RDDT. As described in the Preliminary Studies section, previous measures of disability were used for persons in long term care (LTC) and thus, need to be validated for use in the ED. The retrospective analysis will determine which indicators have superior measurement properties for use in the ED, plus, the retrospective analyses will link ED patient disability to health outcomes a necessary external validation step. A modified RDDT will be used in the prospective phase of the study. As lengthy diagnostic tools are neither feasible nor practical in the ED, Rasch scales are more useful in that subsets scale well and retain their measurement properties that remain accurate and precise. The investigators will conduct a randomized clinical trial (prospective phase) allocating patients into the study arm utilizing the RDDT (new tool) to compare with the control arm (standard care using MOD) to determine which measure is more accurate and precise as a measure of disability. There are both retrospective and prospective aspects to this multi-methodological interdisciplinary study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the adult ED at the Yale New Haven Hospital (YNHH)
* 65 years or older
* Medicare recipients
* Community dwellers.

Exclusion Criteria:

* Patients and their guardians will be excluded for the following reasons:

  1. Non English speaking
  2. suffering from a condition that precludes interview i.e. communication impairment
  3. unable to provide two contact numbers for follow-up
  4. presenting with acute psychosis or are suicidal.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 635 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the presence/absence of at least one visit to the ED, hospital admission or death within 90 days of the initial ED visit. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Post, PhD, Principal Investigator — Yale University School of Medicine, Emergency Medicine
Locations (2):
- United States (2):
  - Yale New Haven Emergency Department, New Haven, Connecticut
  - Yale University, Emergency Department, New Haven, Connecticut

REFERENCES:
- [Background] Post LA, Salmon CT, Prokhorov A, Oehmke J, Swierenga SJ. Aging and elder abuse: Projections for Michigan. In: Murdock SH, Swanson DA, eds. Applied Demography in the 21st Century: Springer Publications; 2008.
- [Background] Post LA, Swierenga SJ, Oehmke J, et al. The implications of an aging population structure. International Journal of the Interdisciplinary Social Sciences. 2006;1(2):47-57.
- [Background] Bodenheimer T, Fernandez A. High and rising health care costs. Part 4: can costs be controlled while preserving quality? Ann Intern Med. 2005 Jul 5;143(1):26-31. doi: 10.7326/0003-4819-143-1-200507050-00007. PMID 15998752
- [Background] Oehmke J, Tsukamati, Post LA. Can health care services attract retirees and contribute to the economic stability of rural places? Agriculture and Resource Economics Review. 2007;36(1):95-106.
- [Background] Cunningham PJ. Medicaid/SCHIP cuts and hospital emergency department use. Health Aff (Millwood). 2006 Jan-Feb;25(1):237-47. doi: 10.1377/hlthaff.25.1.237. PMID 16403760
- [Background] Cunningham PJ. What accounts for differences in the use of hospital emergency departments across U.S. communities? Health Aff (Millwood). 2006 Sep-Oct;25(5):w324-36. doi: 10.1377/hlthaff.25.w324. Epub 2006 Jul 18. PMID 16849363
- [Background] Wharam JF, Landon BE, Galbraith AA, Kleinman KP, Soumerai SB, Ross-Degnan D. Emergency department use and subsequent hospitalizations among members of a high-deductible health plan. JAMA. 2007 Mar 14;297(10):1093-102. doi: 10.1001/jama.297.10.1093. PMID 17356030
- [Background] McCaig LF, Xu J, Niska RW. Centers for Disease Control and Prevention. Estimates of Emergency Department Capacity: United States, 2007. NCHS Health E-Stat [http://www.cdc.gov/nchs/data/hestat/ed_capacity/ED_capacity.htm. Accessed October 21, 2009, 2009.
- [Background] AHRQ. National Healthcare Quality Report 2008: March 2009 2009. 09-0001.Accessed www.ahrq.gov/qual/qrdr08.htm
- [Background] Oliver D, Connelly JB, Victor CR, Shaw FE, Whitehead A, Genc Y, Vanoli A, Martin FC, Gosney MA. Strategies to prevent falls and fractures in hospitals and care homes and effect of cognitive impairment: systematic review and meta-analyses. BMJ. 2007 Jan 13;334(7584):82. doi: 10.1136/bmj.39049.706493.55. Epub 2006 Dec 8. PMID 17158580
- [Background] Chelly JEMDPMBA, Conroy LRNMSNMPM, Miller GAS, Elliott MNP, Horne JLBA, Hudson MEMD. Risk Factors and Injury Associated With Falls in Elderly Hospitalized Patients in a Community Hospital. Journal of Patient Safety. 2008;4(3):178-183.
- [Background] Harbarth S, Fankhauser C, Schrenzel J, Christenson J, Gervaz P, Bandiera-Clerc C, Renzi G, Vernaz N, Sax H, Pittet D. Universal screening for methicillin-resistant Staphylococcus aureus at hospital admission and nosocomial infection in surgical patients. JAMA. 2008 Mar 12;299(10):1149-57. doi: 10.1001/jama.299.10.1149. PMID 18334690
- [Background] Rodriguez-Molinero A, Lopez-Dieguez M, Tabuenca AI, de la Cruz JJ, Banegas JR. Functional assessment of older patients in the emergency department: comparison between standard instruments, medical records and physicians' perceptions. BMC Geriatr. 2006 Sep 4;6:13. doi: 10.1186/1471-2318-6-13. PMID 16952319
- [Background] Peikes D, Chen A, Schore J, Brown R. Effects of care coordination on hospitalization, quality of care, and health care expenditures among Medicare beneficiaries: 15 randomized trials. JAMA. 2009 Feb 11;301(6):603-18. doi: 10.1001/jama.2009.126. PMID 19211468
- [Background] Jack BW, Chetty VK, Anthony D, Greenwald JL, Sanchez GM, Johnson AE, Forsythe SR, O'Donnell JK, Paasche-Orlow MK, Manasseh C, Martin S, Culpepper L. A reengineered hospital discharge program to decrease rehospitalization: a randomized trial. Ann Intern Med. 2009 Feb 3;150(3):178-87. doi: 10.7326/0003-4819-150-3-200902030-00007. PMID 19189907
- [Background] Clancy CM. Reengineering hospital discharge: a protocol to improve patient safety, reduce costs, and boost patient satisfaction. Am J Med Qual. 2009 Jul-Aug;24(4):344-6. doi: 10.1177/1062860609338131. Epub 2009 Jun 5. No abstract available. PMID 19502567
- [Background] Epstein AM. Revisiting readmissions--changing the incentives for shared accountability. N Engl J Med. 2009 Apr 2;360(14):1457-9. doi: 10.1056/NEJMe0901006. No abstract available. PMID 19339727
- [Background] Mion LC, Palmer RM, Meldon SW, Bass DM, Singer ME, Payne SM, Lewicki LJ, Drew BL, Connor JT, Campbell JW, Emerman C. Case finding and referral model for emergency department elders: a randomized clinical trial. Ann Emerg Med. 2003 Jan;41(1):57-68. doi: 10.1067/mem.2003.3. PMID 12514683
- [Background] Strange GR, Chen EH. Use of emergency departments by elder patients: a five-year follow-up study. Acad Emerg Med. 1998 Dec;5(12):1157-62. doi: 10.1111/j.1553-2712.1998.tb02688.x. PMID 9864128
- [Background] McCaig LF, Nawar EW. National Hospital Ambulatory Medical Care Survey: 2004 emergency department summary. Adv Data. 2006 Jun 23;(372):1-29. PMID 16841785
- [Background] Cooke MW, Arora P, Mason S. Discharge from triage: modelling the potential in different types of emergency department. Emerg Med J. 2003 Mar;20(2):131-3. doi: 10.1136/emj.20.2.131. PMID 12642524
- [Background] Conner T, Prokhorov A, Page C, Fang Y, Xiao Y, Post LA. Impairment and abuse of elderly by staff in long-term care in Michigan: evidence from structural equation modeling. J Interpers Violence. 2011 Jan;26(1):21-33. doi: 10.1177/0886260510362880. Epub 2010 May 6. PMID 20448233
- [Background] Hahn EA, Cella D. Health outcomes assessment in vulnerable populations: measurement challenges and recommendations. Arch Phys Med Rehabil. 2003 Apr;84(4 Suppl 2):S35-42. doi: 10.1053/apmr.2003.50245. PMID 12692770
- [Background] Stiell A, Forster AJ, Stiell IG, van Walraven C. Prevalence of information gaps in the emergency department and the effect on patient outcomes. CMAJ. 2003 Nov 11;169(10):1023-8. PMID 14609971
- [Background] Caplan GA, Williams AJ, Daly B, Abraham K. A randomized, controlled trial of comprehensive geriatric assessment and multidisciplinary intervention after discharge of elderly from the emergency department--the DEED II study. J Am Geriatr Soc. 2004 Sep;52(9):1417-23. doi: 10.1111/j.1532-5415.2004.52401.x. PMID 15341540
- [Background] Osborne JW. Best Practices in Quantitative Methods. Thousand Oaks, CA: Sage Publications, Inc.; 2008.
- [Background] Hustey FM, Mion LC, Connor JT, Emerman CL, Campbell J, Palmer RM. A brief risk stratification tool to predict functional decline in older adults discharged from emergency departments. J Am Geriatr Soc. 2007 Aug;55(8):1269-74. doi: 10.1111/j.1532-5415.2007.01272.x. PMID 17661968
- [Background] Peterson PG. The shape of things to come: Global aging in the twenty-first century. Journal of International Affairs. 2002;56(1):189-210.
- [Background] Post LA, Fulk R, Biroscak BJ. Violence prevention informatic systems. The International Journal of Technology, Knowledge and Society. 2008;4(2):155-162.
- [Background] Taeuber C. US Department of Commerce, Economics, and Statistics Administration, Bureau of the Census. Sixty-five plus in America. Current population reports. Special studies. Washington, DC 1996. P23-173RV.Accessed
- [Background] National Center for Health Statistics (US). Health, United States, 2007: With Chartbook on Trends in the Health of Americans. Hyattsville (MD): National Center for Health Statistics (US); 2007 Nov. Report No.: 2007-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK21014/ PMID 20698068
- [Background] Miller T. Increasing longevity and Medicare expenditures. Demography. 2001 May;38(2):215-26. doi: 10.1353/dem.2001.0018. PMID 11392909
- [Background] Covinsky KE, Palmer RM, Fortinsky RH, Counsell SR, Stewart AL, Kresevic D, Burant CJ, Landefeld CS. Loss of independence in activities of daily living in older adults hospitalized with medical illnesses: increased vulnerability with age. J Am Geriatr Soc. 2003 Apr;51(4):451-8. doi: 10.1046/j.1532-5415.2003.51152.x. PMID 12657063
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] Caplan GA, Brown A, Croker WD, Doolan J. Risk of admission within 4 weeks of discharge of elderly patients from the emergency department--the DEED study. Discharge of elderly from emergency department. Age Ageing. 1998 Nov;27(6):697-702. doi: 10.1093/ageing/27.6.697. PMID 10408663
- [Background] Currie CT, Lawson PM, Robertson CE, Jones A. Elderly patients discharged from an accident and emergency department--their dependency and support. Arch Emerg Med. 1984 Dec;1(4):205-13. doi: 10.1136/emj.1.4.205. PMID 6100354
- [Background] McCusker J, Verdon J, Tousignant P, de Courval LP, Dendukuri N, Belzile E. Rapid emergency department intervention for older people reduces risk of functional decline: results of a multicenter randomized trial. J Am Geriatr Soc. 2001 Oct;49(10):1272-81. doi: 10.1046/j.1532-5415.2001.49254.x. PMID 11890484
- [Background] Callahan EH, Thomas DC, Goldhirsch SL, Leipzig RM. Geriatric hospital medicine. Med Clin North Am. 2002 Jul;86(4):707-29. doi: 10.1016/s0025-7125(02)00014-7. PMID 12365337